CLINICAL TRIAL: NCT02100059
Title: Motor and Sensory Deficits Following Partial Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-16795
Record Dates: First submitted 2014-01-13; First posted 2014-03-31 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Meniscus Tear
Keywords: meniscectomy; arthroscopic partial meniscectomy; meniscus
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical Stimulation (TENS) (Experimental): The TENS (transcutaneous electrical nerve stimulation) electrodes will be applied on the medial and lateral superior, as well as the medial and lateral inferior, borders of the patella. A continuous biphasic pulsatile current (150 Hz, phase duration 150 µs) will be applied at an intensity that produces a comfortable sensation but not a muscle contraction. The duration of intervention will be 40 minutes.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation — The TENS electrodes will be applied on the medial and lateral superior, as well as the medial and lateral inferior, borders of the patella. A continuous biphasic pulsatile current (150 Hz, phase duration 150 µs) will be applied at an intensity that produces a comfortable sensation but not a muscle contraction. The duration of intervention will be 40 minutes.
  Other Names: TENS; Sensory TENS

SUMMARY:
To determine changes in thigh muscle function and knee pain after a partial meniscectomy surgery and to also determine the effects of applying electrical stimulation to the knee to determine if this improves thigh muscle function and decreases pain.

DETAILED DESCRIPTION:
The objective for this study is to determine the differences in corticospinal excitability and central sensitization of nociceptive pathways in individuals with a history of arthroscopic partial meniscectomy compared to healthy controls. Our central hypothesis is that quadriceps weakness following partial meniscectomy is due to higher levels of corticospinal excitability and central sensitization of nociceptive pathways, which can be modified with therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-65
* Arthroscopic partial meniscectomy with in the past 15 years

Exclusion Criteria:

* History of traumatic spine or lower extremity injury within the last 6 months
* Previous adverse reaction to electrical stimulation (i.e. burns or hypersensitivity)
* Cardiac pacemaker
* Metal implants in head
* Current pregnancy
* Neurological disorders
* History of seizures
* Unable to give consent or understand the procedures of this study

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in quadriceps force output and voluntary activation | Single Study Visit
  Quadriceps activation will be estimated by utilizing the burst-superimposition technique on a maximum voluntary isometric contraction (MVIC) and during a resting condition.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ACT, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States